CLINICAL TRIAL: NCT04803162
Title: The Role of High-resolution Esophageal Manometry and Specific Biomarkers of Inflammation in the Diagnosis of Patients With Dysphagia and Suspected Eosinophilic Esophagitis
Brief Title: The Role of HRM and Specific Biomarkers of Inflammation in the Diagnosis of Patients With Dysphagia and Suspected EoE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Sarbinowska, MD, Wroclaw Medical University
Other Study IDs: STM.C130.17.045
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Eosinophilic Esophagitis
Keywords: eosinophilic esophagitis; eotaxin 3; major basic protein; interleukin 5; interleukin 13; transforming growth factor beta 1; high-resolution manometry; Gastrointestinal Quality of Life index
MeSH Terms: conditions — Eosinophilic Esophagitis; Rhinitis, Allergic; Camurati-Engelmann Syndrome | interventions — Omeprazole; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fixed tissue, serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with eosinophilic esophagitis: Each project participant completed a health and existing disease questionnaire and the GIQLI. Quantification of IL-5, IL-13 and TGF-β1 serum levels was performed using enzyme immunoassays. From each participant during the esophagogastroduodenoscopy, 6 oesophageal mucosa biopsy specimens were collected. The obtained material was sent for histopathological examination to assess peak eosinophil count (PEC). After completing medical examinations, the project participants were divided according to the histopathological criterion's fulfillment for the diagnosis of EoE. Patients with ≥15 eosinophils/HPF in the biopsy samples constituted the group of patients with EoE, while the remaining patients - the control group. EoE patients were then treated for 8 weeks with PPs - omeprazole in the dose of 20 mg twice daily. After 8 weeks, each patient in the EoE group again passed all the tests (the protocols were identical to those used for qualifying patients to the project).
  Interventions: Diagnostic Test: High-resolution manometry; Diagnostic Test: Serum biomarkers; Diagnostic Test: Gastrointestinal Quality of Life index; Drug: Omeprazole 20 MG Oral Tablet
- patients without eosinophilic esophagitis: Each project participant completed a health and existing disease questionnaire and the GIQLI. Quantification of IL-5, IL-13 and TGF-β1 serum levels was performed using enzyme immunoassays. From each participant during the esophagogastroduodenoscopy, 6 oesophageal mucosa biopsy specimens were collected. The obtained material was sent for histopathological examination to assess peak eosinophil count (PEC). After completing medical examinations, the project participants were divided according to the histopathological criterion's fulfillment for the diagnosis of EoE. Patients with ≥15 eosinophils/HPF in the biopsy samples constituted the group of patients with EoE, while the remaining patients - the control group.
  Interventions: Diagnostic Test: High-resolution manometry; Diagnostic Test: Serum biomarkers; Diagnostic Test: Gastrointestinal Quality of Life index

INTERVENTIONS:
Diagnostic Test: High-resolution manometry — The parameters of high-resolution esophageal manometry will be compared between EoE patients and controls.
Diagnostic Test: Serum biomarkers — The serum levels of IL-5, IL-13, TGF-β1, MBP and eotaxin 3 will be compared between EoE patients and controls.
Diagnostic Test: Gastrointestinal Quality of Life index — The Gastrointestinal Quality of Life index (GIQLI) will be compared between EoE patients and controls.
Drug: Omeprazole 20 MG Oral Tablet — The parameters of high-resolution esophageal manometry and serum levels of IL-5, IL-13, TGF-β1, MBP and eotaxin 3 will be compared in the group of patients with EoE at enrollment in the project and after 3 months of treatment with PPIs.
  Other Names: Omeprazole in the dose of 20 mg twice daily
  Groups: patients with eosinophilic esophagitis

SUMMARY:
The aim of the project is to assess the correlation between the results of high-resolution oesophageal manometry and specific biomarkers of inflammation (eotaxin 3, major basic protein, IL-5, IL-13, TGF-beta1) with symptoms of dysphagia, endoscopic and histological features and the assessment of quality of life in patients with eosinophilic esophagitis.

Research hypothesis: The results of high resolution esophageal manometry (HRM) and specific inflammatory biomarkers correlate with symptoms of dysphagia, endoscopic and histological features, and assessment of quality of life in patients with eosinophilic oesophagitis. HRM, along with the determination of specific inflammatory biomarkers present in the peripheral blood, may serve as a less invasive method of assessing the effectiveness of the treatment of eosinophilic oesophagitis in relation to the currently used endoscopic examinations.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age,
* patients referred for endoscopic diagnostics due to dysphagia.

Exclusion Criteria:

* already diagnosed chronic diseases with possible eosinophilic infiltration of the gastrointestinal tract (eosinophilic esophagitis, eosinophilic gastroenteritis, Crohn's disease, celiac disease),
* rheumatological, dermatological and genetic disorders with possible peripheral eosinophilia,
* dysphagia caused by a diagnosed neoplastic infiltration of the esophagus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at the Department of Gastroenterology and Hepatology and the Department of Otolaryngology, Head and Neck Surgery at Wroclaw Medical University in Poland from 1.11.2017 to 31.12.2021 for endoscopic diagnosis of dysphagia.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
High-resolution manometry | 3 months
  The parameters of high-resolution esophageal manometry will be compared between EoE patients and controls.
Serum biomarkers | 3 months
  The serum levels of IL-5, IL-13, TGF-β1, MBP and eotaxin 3 will be compared between EoE patients and controls.
Gastrointestinal Quality of Life index | 3 months
  The Gastrointestinal Quality of Life index (GIQLI) will be compared between EoE patients and controls.

SECONDARY OUTCOMES:
High-resolution manometry in the group of patients with EoE | 3 months
  The parameters of high-resolution esophageal manometry will be compared in the group of patients with EoE at enrollment in the project and after 3 months of treatment with PPIs.
Serum biomarkers in the group of patients with EoE | 3 months
  The serum levels of IL-5, IL-13, TGF-β1, MBP and eotaxin 3 will be compared in the group of patients with EoE at enrollment in the project and after 3 months of treatment with PPIs.

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Waśko-Czopnik, PhD MD, Principal Investigator — Department of Gastroenterology and Hepatology, Wroclaw Medical University
Locations (1):
- Department of Gastroenterology and Hepatology, Wroclaw Medical University, Wroclaw, Borowska 213, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarbinowska J, Wiatrak B, Wasko-Czopnik D. Esophageal Motility Disorders in the Natural History of Acid-Dependent Causes of Dysphagia and Their Influence on Patients' Quality of Life-A Prospective Cohort Study. Int J Environ Res Public Health. 2021 Oct 23;18(21):11138. doi: 10.3390/ijerph182111138. PMID 34769657